CLINICAL TRIAL: NCT00425698
Title: Effect of Erythropoietin on Renal Function After Kidney Transplantation
Brief Title: Erythropoietin (EPO) and Ischemia-reperfusion After Kidney Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Danilo Fliser, MD, Professor of Medicine, Saarland University Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MHH - EPONTX - 01/06
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous erythropoietin (Active Comparator): Erythropoietin alpha 3 x 40.000 IU intraarterial or intravenous within 7 days after cadaveric kidney transplantation
  Interventions: Drug: Recombinant erythropoietin alpha (rHuEPO alpha); Drug: Placebo
- intravenous placebo (Placebo Comparator): Placebo 3x IU intraarterial or intravenous within 7 days after cadaveric kidney transplantation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant erythropoietin alpha (rHuEPO alpha) — Erythropoietin alpha 3 x 40.000 IU intraarterial or intravenous within 7 days after cadaveric kidney transplantation
  Other Names: Erypo
  Arms: intravenous erythropoietin
Drug: Placebo — Placebo 3x IU intraarterial or intravenous within 7 days after cadaveric kidney transplantation

SUMMARY:
The hematopoetic cytokine erythropoietin (EPO) has been shown to reduce programmed cell death and tissue destruction in experimental models of acute kidney ischemia-reperfusion injury. Thus, treatment with high dose recombinant human EPO (rHuEPO) may prevent kidney tissue damage and loss of renal function after successful kidney transplantation in humans.

DETAILED DESCRIPTION:
Erythropoietin (EPO) has pleiotropic effects well beyond the maintenance of red blood cell mass. In the embryo, EPO is a major regulator of vascular formation and organ growth, and EPO receptors are found in almost every embryonic tissue. EPO receptors also exist in many adult tissues including renal tissue, and even the notion of autocrine or paracrine EPO systems has been raised. Although the peritubular fibroblasts are the major adult site for EPO production, EPO receptors have been demonstrated in many kidney cell types, e.g. proximal tubule epithelial cells, mesangial cells, and the glomerulus. Moreover, EPO has important cytoprotective effects on various cell lines and organs, and protection from ischemic injury and inhibition of apoptotic death-related pathways has been reported in brain, heart and renal tissue. The intracellular pathways involved in these favourable EPO effects may involve nuclear translocation of the transcription factor NF- B, JAK2 phosphorylation and phosphorylation of Akt (protein kinase B).

A recent experimental study revealed that cobalt administration to rats caused up-regulation of EPO, and diminished the degree of renal injury caused by ischemia-reperfusion (I/R), suggesting that EPO may also play an important role in renal ischemic preconditioning. Indeed, subsequent studies from different laboratories demonstrated that preconditioning with recombinant human EPO (rHuEPO) is protective against I/R injury in rodents. In this respect data on specific protective effects of rHuEPO and its analogues on endothelial cells of glomeruli are of particular interest. Furthermore, administration of rHuEPO may not have only protective effects on the vascular level, but also potential of regeneration, since EPO also stimulates proliferation and differentiation of regenerative cells such as endothelial progenitor cells (EPCs).

Renal ischemia, whether caused by shock or after surgery, is a major cause of acute renal failure (ARF) in man. In this respect kidney transplantation is a classical model of ARF due to I/R injury, since the transplanted organ is connected to the recipients blood supply usually after several hours of "cold ischemia". Although reperfusion is essential for the survival of ischemic tissue, it also initiates a complex and interrelated sequence of events that results in injury and the eventual death of renal cells as a result of a combination of both apoptosis and necrosis. Apoptotic cell death has been documented in human biopsies after renal I/R, and inhibition of apoptotic signalling and cell death ameliorates the associated injury and inflammation in an experimental model of ischemic ARF. Similarly, I/R damage of transplanted kidney is thought to be a major factor limiting renal function after successful transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female aged 18 to 70 years without restricted legal competence and being able to follow the trial instructions
3. Cadaveric renal transplant, cold ischemia time below 24 h, and standard immunosuppressive regimen
4. A haemoglobin level > 8 and < 14 g/dl
5. Treatment with standard immunosuppression (steroids, cyclosporine A, tacrolimus, MMF or azathioprine)
6. In patient with diabetes mellitus HbA1c < 9%

Exclusion Criteria:

1. Previous or current myelodysplastic or -proliferative disorders
2. History of cancer within the last 5 years.
3. Systemic chemotherapy or radiotherapy
4. Higher degree renal anemia or persistent Hb > 14 g/dl
5. Treatment with other stem cell growth factors cells like GM-CSF, VEGF
6. Bleeding episodes within 3 month prior transplantation
7. Sitting diastolic BP > 110 mmHg or sitting systolic BP > 170 mmHg
8. Known intolerance of rHuEpo or analogs
9. Cardiovascular event within 6 months prior transplantation
10. Thromboembolic event within 6 months prior transplantation
11. Relevant stenosis of extra- and intracranial, and peripheral arteries
12. Systemic diseases (SLE or vasculitis)
13. Acute or chronic infection and/or CRP > 10 mg/l prior transplantation
14. Hemolysis or disorders of blood formation (e.g., thalassemia)
15. Further organ transplants or combined organ transplantation
16. Pregnancy or inadequate contraception
17. Psychiatric or emotional problems, or chronic seizures
18. Unwillingness to participate satisfactorily for the entire trial period
19. Participation in a clinical trial within 30 days prior to study inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danilo Fliser, MD, Principal Investigator — Saarland University Medical Centre
Locations (1):
- Hannover Medical School, Hanover, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2007 until May 2009. Single recruitment site was the Hannover Medical School in Hannover, Germany
Pre-assignment Details: 420 patients screened, 88 patients finally enrolled, other patients not enrolled because of age<18 years, living-related kidney transplantation, high pre-immunisation, multiple transplantation, participation in other studies, no interest for participation or withdraw of consent
Period: Overall Study
Arm/Group | Erythropoietin | Placebo
Started | 44 | 44
Completed | 41 | 42
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin | Placebo | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (2) | 50 (2) | 52 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 25 | 26 | 51
Region of Enrollment [Number; unit: participants]
  Germany | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Kidney Graft Function by Estimated Glomerular Filtration Rate (eGFR)
Description: Estimated glomerular filtration rate (eGFR) was assessed using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration)equation
Time Frame: 42 days after transplantation
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 44 | 44
ml/min | 47 (28) | 46 (22)
Statistical Analysis 1: Comparison: Erythropoietin; Null hypothesis: Erythopoietin significantly improves kidney graft function. Power calculation: with a difference of at least 4 mL/min in mean eGFR between groups the number of patients enrolled per group (at least 41) would allowed the detection of a significant difference between groups at a 5% level (p<0.05); Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 4, Standard Deviation 15

2. Secondary Outcome: Kidney Graft Function by Estimated Glomerular Filtration Rate (eGFR)
Description: as for outcome 1
Time Frame: 6 month after transplantation
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: ml/min

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Erythropoietin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/44 | 1/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin (N=44) | Placebo (N=44)
graft loss (Renal and urinary disorders) | 3 (3) | 0 (0)
embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes